CLINICAL TRIAL: NCT03952819
Title: The Effects of Hemodialysis on Serum Sclerostin Levels in Diabetic Patients With Chronic Renal Failure
Brief Title: The Effects of Hemodialysis on Serum Sclerostin Levels
Acronym: sclerostin
Status: Completed | Type: Observational
Sponsor: Abant Izzet Baysal University (Other)
Responsible Party: Principal Investigator, Ozgur Mehmet Yis, Assist. Prof., Abant Izzet Baysal University
Other Study IDs: AbantIBU-Biochem-OMY-1
Record Dates: First submitted 2019-01-31; First posted 2019-05-16 (Actual); Last update posted 2019-05-16 (Actual); Status verified 2019-05

CONDITIONS: Diabetes Mellitus; Renal Failure; Hemodialysis Access Failure
Keywords: Diabetes Mellitus; Renal Failure; Hemodialysis Access Failure; Sclerostin
MeSH Terms: conditions — Diabetes Mellitus; Renal Insufficiency; Sclerosteosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Diabetic group,: The study was designed with 28 chronic hemodialysis patients (17 men, 11 women) receiving treatment at our hospital. Of the 28 hemodialysis patients, 14 had Type 2 diabetes mellitus. On the day of hemodialysis, blood samples were obtained within 30 minutes of before and after dialysis. Intervention is to take blood samples and determine serum sclerostin level in blood samples. Any drugs or substances will not be given.
  Interventions: Diagnostic Test: serum sclerostin
- Non-Diabetic group,: Of the 28 hemodialysis patients, the other 14 were not diabetic. On the day of hemodialysis, blood samples were obtained within 30 minutes of before and after dialysis. Intervention is to take blood samples and determine serum sclerostin level in blood samples. Any drugs or substances will not be given.
  Interventions: Diagnostic Test: serum sclerostin
- Control group,: The study was designed with 56 individuals; 28 healthy volunteers as a control group. Venous blood samples of the control group were obtained at the blood sampling unit by the healthcare personnel during morning hours following overnight fasting while they were sitting after being rested. The intervention is to take blood samples and determine serum sclerostin level in blood samples. Any drugs or substances will not be given.
  Interventions: Diagnostic Test: serum sclerostin

INTERVENTIONS:
Diagnostic Test: serum sclerostin — blood samples obtained

SUMMARY:
Background: Parathyroid hormone (PTH) and 1,25-dihydroxy vitamin D (1,25-OHD) as well as mineral bone metabolism modulators like sclerostin are thought to play an important role in in diabetic patients with chronic renal failure. The present study aimed to analyse the levels of serum sclerostin before and after hemodialysis which is a primary element of treatment in such combined disease states.

Methods: Serum sclerostin concentrations were measured using a commercially available enzyme-linked immunosorbent assay kit with 56 individuals who 14 chronic hemodialysis patients with diabetes, 14 chronic hemodialysis patients with non-diabetes and 28 healthy volunteers as a control group.

DETAILED DESCRIPTION:
Sclerostin results in a phenotype characterized by high bone mass (sclerosteosis) in humans, it is produced by osteocytes and chondrocytes, it suppresses osteoblast activity by inhibiting canonicular Wnt / β-catenin signal, it is described as an anti-anabolic protein of 22-kDa size.In diabetes mellitus patients osteoporosis and obesity always create problems, increased levels of sclerostin inhibit canonicular Wnt / β-catenin signal and is potentially held responsible from bone fragility. Bone problems are important both for chronic kidney disease patients and diabetes mellitus patients and in instances where these two diseases coexist, the importance of sclerostin as a new marker of bone turnover increases. The objective of this study is to evaluate how serum sclerostin levels are affected in diabetes mellitus patients undergoing hemodialysis treatment. To this end, the investigators analyzed the levels of serum sclerostin before and after hemodialysis as it is a main element of treatment in such combined disease states.

ELIGIBILITY:
Inclusion Criteria:

* Patients who satisfied inclusion criteria signed informed consent forms before they enrolled in the study.
* Chronic hemodialysis patients receiving treatment at our hospital.
* The patients had Type 2 diabetes mellitus and the patients were not diabetic.
* Healthy volunteers as a control group

Exclusion Criteria:

* Clinical diagnosis of chronic respiratory failure, acute kidney failure, nephrotic syndrome, end-stage liver disease, malignancy, acute infections
* Any health problems necessitating urgent interventions, drinking alcohol and/or smoking as well as pregnant patients

Ages: 44 Years to 74 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study was designed with 56 individuals; 28 chronic hemodialysis patients (17 men, 11 women) receiving treatment at our hospital and 28 healthy volunteers as a control group. Of the 28 hemodialysis patients, 14 had Type 2 diabetes mellitus while the other 14 were not diabetic.
Sampling Method: Probability Sample
Enrollment: 56 (Actual)
Dates: Start 2017-09-14 (Actual); Primary Completion 2018-11-15 (Actual); Study Completion 2018-12-15 (Actual)

PRIMARY OUTCOMES:
change from levels of serum sclerostin of Diabetic group in dialysis at 1 months | blood samples were obtained within 30 minutes of before and after dialysis
  Sclerostin is an anti-anabolic protein of 22-kDa size, at a level of ng/mL. Serum concentrations are measured with an ELISA kit (Cloud-CloneCorp., Katy, TX 77494, USA).
change from levels of serum sclerostin of Non-diabetic group in dialysis at 1 months | blood samples were obtained within 30 minutes of before and after dialysis
  Sclerostin is an anti-anabolic protein of 22-kDa size, at a level of ng/mL. Serum concentrations are measured with an ELISA kit (Cloud-CloneCorp., Katy, TX 77494, USA).
change from levels of serum sclerostin of control group | through study completion, an average of 1 day.
  Sclerostin is an anti-anabolic protein of 22-kDa size, at a level of ng/mL. Serum concentrations are measured with an ELISA kit (Cloud-CloneCorp., Katy, TX 77494, USA).

CONTACTS AND LOCATIONS:
Overall Officials: Ozgur M. Yis, Study Director — BAİBÜ
Locations (1):
- Bolu Abant Izzet Baysal University, Bolu, Merkez, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No